CLINICAL TRIAL: NCT01370733
Title: Evaluation of Low Emission NeoSync EEG Synchronized TMS Technology for the Treatment of Major Depressive Disorder: A Multicenter, Randomized, Double-Blind, Sham-Controlled, Trial
Brief Title: Synchronized Transcranial Magnetic Stimulation (sTMS) in Major Depressive Disorder
Acronym: NEST-MDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NND3001
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Major Depressive Disorder
Keywords: TMS,; MDD,; Depression,; sTMS,; NEST,; NeoSync,; EEG,; synchronous,; non-invasive neuromodulation,; transcranial magnetic stimulation,; antidepressant,
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active sTMS (Experimental): Treatment with the NEST-1 Device
  Interventions: Device: NEST-1 (NeoSync EEG Synchronized TMS)
- Sham (Sham Comparator): Treatment with a sham (inactive) device, identical in sound and appearance to the NEST-1 Device
  Interventions: Device: SHAM

INTERVENTIONS:
Device: NEST-1 (NeoSync EEG Synchronized TMS) — The NeoSync EEG Synchronized TMS (NEST) is an electromechanical medical device that produces and delivers a sinusoidal magnetic field to areas of the brain in the treatment of Major Depressive Disorder.
  Arms: Active sTMS
Device: SHAM — The sham device is configured to simulate the actual NEST-1 device without sTMS therapy being actively delivered.
  Arms: Sham

SUMMARY:
This study is designed to evaluate the safety and efficacy of synchronized transcranial magnetic stimulation (sTMS) using the NeoSync EEG Synchronized TMS device (NEST) in subjects with Major Depressive Disorder. This is a multicenter study in which subjects will be randomized to receive treatment 5 days per week for 6 weeks. Subjects who complete 6 weeks of double-blind treatment may be eligible to receive up to four weeks of open label sTMS therapy or antidepressant medications during the follow-up phase of the study. Follow-up evaluation visits will be conducted during those four weeks, with the frequency of the visits determined by the treatment choice during that timeframe.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a mental disorder associated with significant functional impairment and disability. Affected individuals present with depressed mood, loss of interest or pleasure, feelings of guilt, low self-worth, disturbed sleep or appetite, low energy, and poor concentration.

Psychopharmacological therapy as today's mainstream treatment has revolutionized the clinical management for major depressive disorders and has been shown to improve the quality of life for many patients. With that, these therapies are not effective for all patients. Results released from the Sequenced Treatment Alternatives to Relieve Depression Study (STAR*D), conducted by the National Institute of Mental Health (NIMH), show that approximately 30% of depressed subjects respond to an SSRI in their first trial, despite adequate dosing and duration of treatment. The SSRI antidepressants do have a more favorable side effect profile than older medications, but they still may be difficult for some patients to tolerate because of gastrointestinal distress, anxiety, insomnia, and sexual dysfunction.

In addition to the psychopharmacologic treatments for depression, other therapies such as electroconvulsive therapy (ECT) and repetitive transcranial magnetic stimulation (rTMS) have been shown to have a therapeutic effect in MDD. ECT induces seizures electrically in anesthetized subjects. It is generally safe and effective; however the procedure can have the negative side effect of memory loss and confusion. Treatment with repetitive stimulation (rTMS) is intended to stimulate groups of cells in areas of the brain linked to MDD. While the therapy is non-invasive, it is expensive, involves a complex method for locating the point of stimulation in the brain, and has the potential for seizures.

rTMS uses magnetic pulses which causes neuronal activation of specific areas in the brain. It is generally believed that this activation causes resetting of cortical oscillators to create a therapeutic effect in MDD. The investigators hypothesize that TMS using low energy, sinusoidal magnetic fields synchronized to a patient's individual alpha frequency,(sTMS), can also affect neuronal activity leading to a reemergence of intrinsic rhythms and clinical improvement in MDD. Preliminary study results using sTMS have shown improvements in depressive symptoms with minimal side effects.

This multicenter study is designed to evaluate the safety and efficacy of sTMS in subjects with Major Depressive Disorder. Subjects will be randomized to receive treatment 5 days per week for 6 weeks. At the end of Treatment Week 6, subject will have completed the study treatments and will be offered open label sTMS therapy or alternate antidepressant treatment as clinically indicated. At minimum, subjects will be asked to return for one follow-up visit four weeks after their last double-blind treatment (Week 10) for evaluation and study completion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet the DSM-IV-TR primary diagnosis of initial or recurrent Major Depressive Disorder by DSM-IV-TR criteria rendered by structured interview using the Mini International Neuropsychiatric Interview (MINI).
* HAM-D17 score >= 17 and Item 1 score greater than or equal to 2.
* Duration of current episode >=8 weeks. The definition of an episode is demarcated by a period of >=2 months when the subject did not meet full criteria for the DSM-IV-TR definition of Major Depressive Episode. Maximum duration of current episode cannot exceed 2 years.
* The baseline EEG is of sufficient duration and quality that it can be processed for quantitative analysis.
* Subjects are willing and able to adhere to the intensive treatment schedule and all required study visits.

Exclusion Criteria:

* Subjects are unable or unwilling to give informed consent.
* Diagnosed with the following conditions (current unless otherwise stated):

  * Any other current primary Axis I mood, anxiety, or psychotic disorder, including bipolar disorder.
  * Depression secondary to a general medical condition, or substance-induced.
  * History of substance abuse or dependence within the past 6 months (except nicotine and caffeine).
  * Any bipolar disorder or psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features in this or previous episodes.
  * Eating disorder (current or within the past year).
  * Obsessive compulsive disorder (lifetime).
  * Post-traumatic stress disorder (current or within the past year).
  * ADHD (currently being treated).
* Subjects meeting criteria for Axis II cluster A or B diagnosis based upon DSM-IV TR criteria, which in the judgment of the Investigator may hinder the subjects in completing the procedures required by the study protocol.
* Subjects with a clinically defined neurological disorder including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure.
  * Space occupying brain lesion.
  * Any history of seizure EXCEPT those therapeutically induced by ECT (childhood febrile seizures are acceptable and these subjects may be included in the study).
  * History of stroke.
  * Transient ischemic attack within two years.
  * Cerebral aneurysm.
  * Dementia.
  * Mini Mental Status Exam (MMSE-2) score of =<24.
  * Parkinson's disease.
  * Huntington's disease.
  * Multiple sclerosis.
  * Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or currently taking medication that lowers the seizure threshold. Medications that lower the seizure threshold are included in the Prohibited Concomitant Medication (Section 5.7).
* Subjects who are currently hospitalized due to severity of depression symptoms.
* Subjects with any of the following treatment histories:

  * TMS treatment within 6 months prior to the screening visit.
  * ECT treatment within 1 year prior to the screening visit.
  * Failure to respond to TMS or ECT treatment (i.e., consistent with ATHF confidence level 3 or higher) in this or any previous episode.
  * Lifetime history of treatment with Deep Brain Stimulation or Vagus Nerve Stimulation.
  * Use of any investigational drug or device within 4 weeks of the randomization visit.
  * Subjects who have been treated with fluoxetine within the past four weeks.
  * If participating in psychotherapy, must have been in stable treatment for at least 2 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the trial.
  * Failure to respond to Monoamine Oxidase Inhibitors (MAOIs) in the current episode.
* Use of any medication(s) listed on the Prohibited Concomitant Medication within 1 week of randomization.
* Subjects are adequately benefiting from current antidepressant medication(s).
* Significant acute suicide risk, defined as:

  * Suicide attempt within the previous 6 months that required medical treatment; or
  * Greater than or equal to 1 suicide attempts in the past 12 months; or
  * Has a clear-cut plan for suicide and states that he/she cannot guarantee that he/she will call his/her regular psychiatrist or the Investigator if the impulse to implement the plan becomes substantial during the study; or
  * In the Investigator's opinion, is likely to attempt suicide within the next 6 months.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
* Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed.
* Clinically significant abnormality or clinically significant unstable medical condition, as indicated by medical history, physical examination, ECG results, or clinical laboratory testing, that in the Investigator's judgment might pose a potential safety risk to the subject or limit interpretation of the trial results, e.g., any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunctioning.
* Women who are currently pregnant or not using a medically acceptable means of birth control and women who are breastfeeding.
* Positive urine drug screen for illicit substances. (A positive urine drug screen at screening may be repeated once prior to randomization).
* Any condition which in the judgment of the Investigator would prevent the subject from completion of the study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Leuchter, MD, Principal Investigator — UCLA Depression Research & Clinic Program
Locations (18):
- United States (18):
  - UCLA Depression Research & Clinic Program, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - UCLA-Harbor, Torrance, California
  - Hartford Hospital Institute of Living, Hartford, Connecticut
  - TMS Specialists Chicago, Chicago, Illinois
  - Sheppard Pratt Health System, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Center for Mood Disorders and Neuromodulation Therapies, UMDNJ-SOM, Cherry Hill, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Brain Stimulation and Neurophysiology Center, Durham, North Carolina
  - Wake Forest University Medical Center, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Mood Disorders Treatment Research Program University of Pittsburgh-Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Butler Hospital Mood Disorders Research Program, Brown Department of Psychiatry and Human Behavior, Providence, Rhode Island
  - MUSC Institute of Psychiatry, Brain Stimulation Lab, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - R/D Clinical Research, Lake Jackson, Texas

REFERENCES:
- [Result] Leuchter AF, Cook IA, Feifel D, Goethe JW, Husain M, Carpenter LL, Thase ME, Krystal AD, Philip NS, Bhati MT, Burke WJ, Howland RH, Sheline YI, Aaronson ST, Iosifescu DV, O'Reardon JP, Gilmer WS, Jain R, Burgoyne KS, Phillips B, Manberg PJ, Massaro J, Hunter AM, Lisanby SH, George MS. Efficacy and Safety of Low-field Synchronized Transcranial Magnetic Stimulation (sTMS) for Treatment of Major Depression. Brain Stimul. 2015 Jul-Aug;8(4):787-94. doi: 10.1016/j.brs.2015.05.005. Epub 2015 May 22. PMID 26143022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred across 17 study sites (both academic and private clinical locations), initiated in May 2012 and all subject visits complete by July 2013. Three sites discontinued early due to departure of the Principal Investigator or due to a loss of contributing staff personnel. None were discontinued specifically due to a lack of enrollment.
Pre-assignment Details: Upon study closure, 291 subjects were consented for possible study participation with 202 of those subjects subsequently enrolled and randomized to treatment. Those entering the study at Screening while currently on an antidepressant required a minimum 1-week wash out period prior to completing a Baseline (Day 0) visit.
Period: Overall Study
Arm/Group | Active sTMS | Sham
Started | 103 | 99
Completed | 86 | 77
Not Completed | 17 | 22
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 3 | 5
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active sTMS | Sham | Total
Number analyzed (Participants) | 103 | 99 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (11.3) | 45.7 (12.2) | 45.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 66 | 128
  Male | 41 | 33 | 74
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian / Alaskan Native | 0 | 2 | 2
  Asian | 5 | 3 | 8
  Black or African American | 6 | 8 | 14
  Hispanic or Latino | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 82 | 79 | 161
  Other or Unknown | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 103 | 99 | 202
Baseline Mean Hamilton Rating Scale for Depression (HAM-D17) [Mean (Standard Deviation); unit: units on a scale] — For this trial, the Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset of the HAM-D28, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials.
  The HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity. A reduction of 50% or more in total score from Baseline indicates clinical response.
  units on a scale | 21.94 (3.46) | 21.15 (3.25) | 21.55 (3.37)
Length of Current Episode in Months [Mean (Standard Deviation); unit: months] | 10.9 (6.8) | 10.8 (6.7) | 10.85 (6.73)
Antidepressant Exposure in Current Episode [Number; unit: participants] — Subjects were asked about previous antidepressant exposure in the current episode. It was possible to select more than one correct response in assessing antidepressant history.
  participants
    Inadequate Dose/Duration of >= 1 Medication | 11 | 13 | 24
    Intolerant of >= 1 Medication | 10 | 5 | 15
    Treatment Naive (ATHF 0) | 40 | 37 | 77
    Adequate Trial of >= 1 Medication | 61 | 65 | 126
Education Level [Number; unit: participants]
  Some high school or less | 2 | 1 | 3
  High school diploma | 19 | 7 | 26
  Vocational school | 1 | 2 | 3
  Some college | 17 | 31 | 48
  College degree | 42 | 42 | 84
  Professional or Graduate degree | 21 | 15 | 36
  Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean HAM-D17 Total Score Change (Intent to Treat - All)
Description: The mean HAM-D17 total score change from Baseline (Day 0) to Week 6 compared between the active treatment and sham-controlled groups. If any subject did not complete the double-blind phase in the ITT population, the assessment last observation carried forward (LOCF) was used. The single value provided in each arm reflects the change seen.
  For this trial, the Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset of the HAM-D28, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. The HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity. A reduction of 50% or more in total score from Baseline indicates clinical response.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Population: Includes all subjects who signed an informed consent, met all I/E criteria, were subsequently randomized and received at least 1 treatment (active sTMS or sham) session in the double-blind phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 103 | 99
units on a scale | -7.49 (7.25) | -6.97 (6.28)

2. Primary Outcome: Mean HAM-D17 Total Score Change (Per Protocol - All)
Description: The mean HAM-D17 total score change from Baseline (Day 0) to Week 6 compared between the active treatment and sham-controlled groups. All subjects in the Per Protocol analysis completed Week 6. Baseline HAM-D17 total score was directly compared to the HAM-D17 total score at Week 6. The single value provided in each arm reflects the change seen.
  For this trial, the Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset of the HAM-D28, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. The HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity. A reduction of 50% or more in total score from Baseline indicates clinical response.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 59 | 61
units on a scale | -9.00 (6.54) | -6.56 (5.85)

3. Secondary Outcome: Mean HAM-D17 Total Score Change (Per Protocol - Non-Naive Subjects)
Description: All subjects in the Per Protocol analysis completed Week 6. Baseline HAM-D17 total score was directly compared to Week 6 HAM-D17 total score. The single value provided in each arm reflects this change.
  This analysis included only Per Protocol subjects exposed to an antidepressant medication in their current episode (non-naive). This includes past history of intolerance, resistance, or inadequate dosing/duration.
  The Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset of the HAM-D28, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. The HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity. A reduction of 50% or more in total score from Baseline indicates clinical response.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Population: Per Protocol Population - Non-Naive Subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 38 | 36
units on a scale | -8.58 (6.93) | -4.25 (4.75)

4. Secondary Outcome: Number of Subjects Who Demonstrate Clinical Response at Week 6 or Early Termination (Intent to Treat)
Description: For this outcome, the Hamilton Rating Scale for Depression (HAM-D17) was utilized to determine clinical response. Response is defined as a reduction of at least 50% in total HAM-D17 score from Baseline through Week 6. If any subject did not complete the double-blind phase (Week 6) in the ITT population, the assessment last observation carried forward (LOCF) was used.
  This outcome provides the total number of subjects in each arm that achieved clinical response within the Intent to Treat population.
  The Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Measure: Number; unit: participants
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 103 | 99
participants | 27 | 25

5. Secondary Outcome: Number of Subjects Who Demonstrate Clinical Response at Week 6 (Per Protocol - All)
Description: For this outcome, the Hamilton Rating Scale for Depression (HAM-D17) was utilized to determine clinical response. Response is defined as a reduction of at least 50% in total HAM-D17 score from Baseline through Week 6. All subjects in the Per Protocol population completed Week 6.
  This outcome provides the total number of subjects in each arm that achieved clinical response within the Per Protocol population.
  The Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 59 | 61
participants | 20 | 18

6. Secondary Outcome: Number of Subjects Who Demonstrate Clinical Response at Week 6 (Per Protocol - Non-Naive Subjects)
Description: The Hamilton Rating Scale for Depression (HAM-D17) was utilized to determine clinical response, defined as a reduction of at least 50% in total HAM-D17 score from Baseline through Week 6. All subjects in the Per Protocol (PP) population completed Week 6. This analysis includes only PP subjects exposed to an antidepressant medication in their current episode (non-naive).
  This outcome provides the total number of subjects in each arm that achieved clinical response within the Non-Naive, Per Protocol population.
  The Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Population: Per Protocol Population - Non-Naive Subjects
Measure: Number; unit: participants
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 38 | 36
participants | 13 | 3

7. Secondary Outcome: Number of Subjects Who Demonstrate Clinical Remission at Week 6 or Early Termination (Intent to Treat)
Description: The Hamilton Rating Scale for Depression (HAM-D17) was utilized to determine clinical remission. Remission is defined as a total HAM-D17 score ≤ 7. If any subject did not complete the double-blind phase (Week 6) in the Intent to Treat (ITT) population, the assessment last observation carried forward (LOCF) was used.
  This outcome provides the total number of subjects in each arm that achieved clinical remission within the ITT population.
  The Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 103 | 99
participants | 11 | 14

8. Secondary Outcome: Number of Subjects Who Demonstrate Clinical Remission at Week 6 (Per Protocol - All)
Description: For this outcome, the Hamilton Rating Scale for Depression (HAM-D17) was utilized to determine clinical remission. Remission is defined as a total HAM-D17 score ≤ 7. All subjects in the Per Protocol population completed Week 6.
  This outcome provides the total number of subjects in each arm that achieved clinical remission within the Per Protocol population at Week 6.
  The Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline to End of Double-Blind Treatment Period (up to week 6)
Population: Per Protocol Population
Measure: Number; unit: participants
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 59 | 61
participants | 9 | 10

9. Secondary Outcome: Number of Subjects Who Demonstrate Clinical Remission at Week 6 or Early Termination (Per Protocol - Non-Naive Subjects)
Description: The Hamilton Rating Scale for Depression (HAM-D17) was utilized to determine clinical remission. Remission is defined as a total HAM-D17 score ≤ 7. All subjects in the Per Protocol population completed Week 6. This analysis includes only PP subjects exposed to an antidepressant medication in their current episode (non-naive).
  This outcome provides the total number of subjects in each arm that achieved clinical remission at Week 6 within the Non-Naive, Per Protocol population.
  The Hamilton Rating Scale for Depression (HAM-D28) was performed as a baseline assessment. A subset, the HAM-D17, was utilized as both a baseline and efficacy measure. It's considered the gold standard for rating depression severity and used frequently in clinical trials. HAM-D17 score ranges from 0-52; a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity.
Time Frame: Baseline to End of Double-Blind Treatment Period (Week 6)
Population: Per Protocol Population - Non-Naive Subjects
Measure: Number; unit: participants
Arm/Group | Active sTMS | Sham
Number analyzed (Participants) | 38 | 36
participants | 5 | 2

ADVERSE EVENTS:
Time Frame: All subject Adverse Events are tracked from the signing of Informed Consent through 4 weeks after the double-blind acute phase has been completed or Early Termination.
Description: Primarily systematic assessments, some reporting was unsolicited although minimal.
Arm/Group | Active sTMS | Sham
Serious Adverse Events (participants affected / at risk) | 2/103 | 1/99
Other Adverse Events (participants affected / at risk) | 80/103 | 42/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active sTMS (N=103) | Sham (N=99)
Hospitalization (Suicide Attempt) (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalization (Risk of Self Harm) (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization (Dehydration) (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active sTMS (N=103) | Sham (N=99)
Tinnitus (Ear and labyrinth disorders) | 3 | 1
Visual Disturbance (Eye disorders) | 3 | 0
Dyschezia (Gastrointestinal disorders) | 3 | 2
Non-Specific GI Discomfort (Gastrointestinal disorders) | 4 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Hand/Arm/Shoulder Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Leg and Foot Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Agitation (Nervous system disorders) | 4 | 1
Dizziness (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 22 | 19
Paresthesia (Nervous system disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 7 | 5
Lack of Energy (Psychiatric disorders) | 3 | 0
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No